CLINICAL TRIAL: NCT00719316
Title: Effect of Aliskiren on Muscle Sympathetic Nerve Activity (MSNA) in Hypertensive Patients With Chronic Kidney Disease
Brief Title: Aliskiren and Muscle Sympathetic Nerve Activity
Acronym: MSNA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Responsible Party: Dr. P. J. Blankestijn, UMC Utrecht
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NL19926.041.07
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2008-07

CONDITIONS: Chronic Kidney Disease; Hypertension; Muscle Sympathetic Nerve Activity
Keywords: Renin inhibitor; Patients; ACE inhibitor or ARB; Chronic Kidney Disease; Hypertension
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension | interventions — aliskiren

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Patients receive Aliskiren 300mg for 6 weeks
  Interventions: Drug: Aliskiren
- Group 2 (No Intervention): 4 weeks no antihypertensive medication

INTERVENTIONS:
Drug: Aliskiren — Aliskiren 300mg per day for 6 weeks
  Other Names: Rasilez 300mg per day
  Arms: Group 1

SUMMARY:
The central hypothesis of this project is that Aliskiren causes a substantial decrease in MSNA in hypertensive patients with CKD.

DETAILED DESCRIPTION:
Cardiovascular (CV) morbidity and mortality are frequently occurring problems in chronic kidney disease (CKD) patients. Apart from the so called traditional risk factors, also risk factors more or less specific to CKD contribute in the pathogenesis of these problems. There is strong evidence that the sympathetic hyperactivity, which often characterizes CKD, is one such factor. Previously, we have shown that angiotensin converting enzyme inhibitors (ACEi) and angiotensin II receptor blockers (ARB) reduce but not normalize this sympathetic hyperactivity. We re-analysed the cohort of patients who were investigated in the past and subsequently treated according to present guidelines. The results show that, despite of treatment, the unfavourable relation between sympathetic hyperactivity and clinical outcome still exits. This might mean that treatment is insufficient. In present study, we want to study the effect of Aliskiren 300mg on sympathetic nerve activity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable chronic kidney disease and hypertension: i.e. using antihypertensive drugs and/or blood pressure > 145/90 mmHg when off medication.
* Patients on ACE inhibitor or ARB

Exclusion Criteria:

* Patients with diabetes mellitus
* Patients on renal replacement therapy
* Pregnant patients Using of antihypertensive which cannot be stopped
* Patients on immunosuppressive therapy and active nephrotic syndrome

Ages: 25 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-07 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Normalisation of muscle sympathetic nerve activity | 1 year

SECONDARY OUTCOMES:
Blood pressure and Blood tests | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: P. J. Blankestijn, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Siddiqi L, Oey PL, Blankestijn PJ. Aliskiren reduces sympathetic nerve activity and blood pressure in chronic kidney disease patients. Nephrol Dial Transplant. 2011 Sep;26(9):2930-4. doi: 10.1093/ndt/gfq857. Epub 2011 Apr 5. PMID 21467128